CLINICAL TRIAL: NCT07298070
Title: Functional and Aesthetic Outcomes Following Lower Lip Reconstruction
Acronym: REFEPLI
Status: Not yet recruiting | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD1425; 2025-A01933-46 (Other: ANSM)
Record Dates: First submitted 2025-12-11; First posted 2025-12-23 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Lower Lip Tissue Loss; Cancer
Keywords: Aesthetic and functional outcomes after lower lip reconstruction; Patient-reported outcome questionnaire; Post-operative; Aesthetic and functional satisfaction; Quality of life; Optimal patient care; Analysis of physicians and surgeons working on topics related to the face
MeSH Terms: conditions — Neoplasms | interventions — Postoperative Period

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patient-Reported Outcome Questionnaire (post-operative) — The patient must complete two questionnaires to assess the functional and aesthetic outcomes and quality of life after lower lip reconstruction. No intervention was assigned by the investigator; the surgery was part of routine clinical care.

SUMMARY:
This retrospective study, aims to evaluate the functional and aesthetic results of lower lip reconstructions, incorporating both patient experiences and the analysis of physicians and surgeons working on facial issues (plastic surgeons and dermatologists) in order to optimize future therapeutic strategies.

DETAILED DESCRIPTION:
Most lip tissue loss is secondary to cancer resection, but other causes may be responsible for this loss, whether in the upper or lower lip: trauma, infectious diseases, giant congenital nevi, hemangiomas, or clefts (labial or cleft palate).

Although the overall 5-year survival rate for skin cancers of the lip is 95%, the long-term quality of life of patients remains a major issue. The lip is both a functional and aesthetic unit, essential for speech, articulation, lip competence, eating, and facial expression.

Reconstructing extensive loss of substance in the upper and lower lips remains a surgical challenge due to the complexity of the perioral musculature and soft tissues. Despite significant advances in free transfers, locoregional flaps remain important in subtotal lip reconstruction, offering better tissue and color adaptation, partial preservation of muscle dynamics, and reduced surgical morbidity.

Reconstruction techniques vary depending on the extent of tissue loss. For defects affecting approximately half of the lip, Abbe or Estlander cross flaps using similar tissue allow functional reinnervation within 6 to 12 months. However, use of these techniques is limited by the risk of microstomia. For more extensive tissue loss (exceeding 50% of the lip), advancement or rotation flaps, such as Gilles, Bernard-Webster, or Karapandzic flaps, are preferred. Finally, tissue loss exceeding 80% or extending beyond the labio-mental sulcus or toward the cheek often requires free tissue transfer, with the risk of impaired lip function and a less than optimal aesthetic result.

Historically, the gold standard technique for lower lip reconstruction is that described by Camille Bernard in 1853, modified by Webster in 1960. Although traditionally considered adynamic due to the sectioning of the perioral muscles, clinical experience suggests that preserving the modiolus and its muscular attachments allows for the maintenance of some tone and mobility in the long term. This structure, the point of convergence of the superficial and deep fascias, plays a key role in lip dynamics by connecting the elevators, depressors, and lateral retractors.

A few studies describe facial reconstruction techniques, with the reference for the lower lip being that described by Camille Bernard in 1853, reviewed by Webster in 1960, but few if any of them focus on the functional and aesthetic results after reconstruction. For example, the retrospective analysis conducted by J. Faulhaber's team reports patient satisfaction in terms of aesthetics and function at the usual follow-up appointment, without substantiating the reasons for this alleged satisfaction. In the study conducted by E. E. Ünsal Tuna et al, a questionnaire was developed to collect functional and aesthetic outcomes from patients, but it was completed by healthcare professionals during a follow-up appointment. The same is true in the prospective study conducted by R. Denadai et al, where although patients are asked about their overall satisfaction with the functional aspect of the reconstruction, it is nevertheless healthcare professionals who more accurately assess the functional results after the reconstruction.

This study therefore focuses on analyzing the post-operative experience of patients, as well as gathering the analysis of doctors and surgeons working on facial issues (plastic surgeons and dermatologists). The aim of the study is to optimize future therapeutic strategies by providing factual information to help decide between the various therapeutic options. It is important to ensure optimal patient care, guaranteeing aesthetic and functional satisfaction, combined with an acceptable quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age.
* Patients who underwent lower lip reconstruction after excision for skin carcinoma, operated on in Pontoise between January 1, 2014, and October 31, 2025.
* Patients who had a post-operative follow-up consultation (± 2 months).
* Patients who were informed and did not object to participating in the study

Exclusion Criteria:

* Cognitive impairment preventing completion of the questionnaire.
* Patient under legal protection (guardianship, conservatorship, or judicial protection).
* Patient deceased.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include patients over 18 years of age who underwent lower lip reconstruction after excision for skin carcinoma, operated on in Pontoise between January 1, 2014, and October 31, 2025.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Overall patient satisfaction with the functional and aesthetic outcomes of lip reconstruction at 12 months postoperatively, assessed by a self-reported questionnaire. | 12 months postoperatively (data collected upon return of completed questionnaire)
  On the questionnaire, the patient is asked to rate from 1 to 10, where 1 means "strongly disagree" and 10 means "strongly agree."

SECONDARY OUTCOMES:
Correlation between overall patient satisfaction and various functional and aesthetic aspects of the face and their impact on daily life. | 12 months postoperatively (data collected upon return of completed questionnaire)
  On the questionnaire, at the end of each subsection, the patient is asked to rate from 1 to 10, where 1 means "strongly disagree" and 10 means "strongly agree."
Postoperative complications up to one year after surgery | Postoperative period from day 0 to one year
  Postoperative complications lasting up to one year, including nonunion, the need for revision surgery, and in particular commissuroplasty.
Quality of life one year after surgery | 12 months postoperatively (data collected upon return of completed questionnaire)
  Quality of Life Questionnaire: University of Washington Quality of Life Questionnaire
Compare patients' aesthetic perceptions with those of professionals | 12 months postoperatively (data collected upon return of completed questionnaire)
  Correlation between aesthetic satisfaction perceived by patients and the one assessed by professionals, using a patient-reported outcome questionnaire and another questionnaire for professionals to evaluate the aesthetic appearance after reconstruction
Demonstrate a correlation between the aesthetic success of the procedure and the technical complexity of its execution. | 12 months postoperatively (data collected upon return of completed questionnaire)
  Evaluation of aesthetic results and technical complexity of procedures based on the technique used, using a questionnaire intended for physicians and surgeons working on topics related to the face

CONTACTS AND LOCATIONS:
Overall Officials: AL TABAA AL TABAA, Dr, Principal Investigator — Hôpital NOVO - Site Pontoise